CLINICAL TRIAL: NCT06488846
Title: Innovative Administration of Long-Acting Injectables for HIV Treatment Enhancement at Home
Acronym: INVITE-Home
Status: Enrolling by invitation | Type: Observational
Sponsor: University of California, San Francisco (Other)
Collaborators: Centers for Disease Control and Prevention (U.S. Federal Agency)
Responsible Party: Sponsor
Other Study IDs: 24-42341; PS005259-02 (Other Grant/Funding Number: Centers for Disease Control and Prevention)
Record Dates: First submitted 2024-06-17; First posted 2024-07-05 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: HIV Infections
Keywords: HIV; Long-acting injectable antiretroviral therapy (LAI-ART)
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Home-Based LAI-ART Administration: People living with HIV receiving LAI-ART in their homes from a trained Treatment Buddy.
  Interventions: Other: INVITE-Home
- Clinic-Based LAI-ART Administration: People living with HIV receiving LAI-ART in clinics from healthcare providers.
  Interventions: Drug: Clinic-Administered LAI-ART
- Oral ART Administration: People living with HIV receiving oral ART medication in clinics from healthcare providers.
  Interventions: Drug: Oral ART

INTERVENTIONS:
Other: INVITE-Home — Curriculum to train Treatment Buddies, selected by the people with HIV, to administer LAI-ART at home with supervision of a Study Nurse.
  Groups: Home-Based LAI-ART Administration
Drug: Clinic-Administered LAI-ART — People with HIV who continue to receive LAI-ART in clinic
  Groups: Clinic-Based LAI-ART Administration
Drug: Oral ART — Oral ART
  Groups: Oral ART Administration

SUMMARY:
This study will support the expansion of long-acting injectable antiretroviral therapy (LAI-ART) in non-clinical settings by developing, implementing, and evaluating a comprehensive, theory-informed training intervention to support the administration of LAI-ART by a trained layperson injector (e.g., friend, family, partner identified by a person living with HIV). This study will address barriers to LAI-ART uptake and persistence, enhance real-world effectiveness, and help close critical HIV care gaps.

DETAILED DESCRIPTION:
There is high interest in long-acting injectable antiretroviral therapy (LAI-ART) among people with (PWH), with many conveniences for uptake and persistence. While LAI-ART eliminate the need for daily pill-taking and have the potential to help close critical gaps in HIV care, patients have expressed important barriers to effective implementation and concerns that frequent clinic visits can exacerbate stigma, increase the risk of unwanted disclosure, and lead to frequent disruptions in their daily lives. The need to travel to a clinic for injection visits multiple times throughout the year can also be financially and logistically prohibitive for many patients and can widen existing healthcare disparities. Similarly, clinicians worry that additional visits outside of routine care may lead to missed appointments, decreased engagement in care, and put further strain on limited clinic resources. Administration of LAI-ART by a trained layperson injector (such as family, friend, or partner of the patient) can help mitigate some of these patient- and clinician-identified barriers. This model of care has been used successfully in other contexts, but up to now it has not been evaluated for HIV treatment. Alternative LAI-ART delivery methods have the potential to increase the PWH and layperson injector's confidence, empowerment, convenience, privacy, and self-management skills, and ultimately facilitate LAI-ART uptake and persistence. INVITE-Home (Innovative Administration of Long-Acting Injectables for HIV Treatment Enhancement at Home) will support the expansion of LAI-ART in non-clinical settings by developing, implementing, and evaluating a comprehensive, theory-informed training to support the administration of LAI-ART by a trained layperson injector. In Aim 1, the investigators will design and develop an innovative, theory-based layperson injector training to improve acceptability and uptake of LAI-ART in home-based settings. Investigators will qualitatively evaluate training barriers and needs of PWH, layperson injectors, and clinicians to develop the training. In Aim 2, investigators will enhance understanding of home-based LAI-ART using the training developed in Phase 1, by examining implementation and effectiveness of home-based LAI-ART injections. This study will address a critical need to develop alternative and decentralized LAI-ART delivery methods that can mitigate barriers to uptake and persistence, enhance the real-world LAI-ART effectiveness, reduce systemic and structural inequities, address clinical and policy challenges, and close key gaps in HIV care.

ELIGIBILITY:
Inclusion Criteria:

PWH:

* Age ≥18 years, patient receiving care at partnering clinical sites;
* can identify a support person injector (i.e., family, friend, or partner) who is willing and able to provide injections;
* has received at least the loading dose of cabotegravir/rilpivirine CAB/RPV (i.e., 600mg/900mg IM) without serious adverse events;
* is virologically suppressed (HIV RNA <50 copies/mL);
* has no history of treatment failure;
* has no known or suspected resistance to either RPV or CAB;
* is interested in receiving home-based injections; is approved by their clinical team as a candidate for home-based injections;
* has the intention to use CAB/RPV for at least 12 months;
* and is willing and able to give informed consent.

Treatment Buddy:

* Age ≥18 years,
* identified by the PWH,
* is willing and able to provide monthly or bimonthly LAI-ART injections at the PWH's place of residence, and
* is willing and able to give informed consent.

Exclusion Criteria:

PWH:

* <18 years of age, not receiving care at partnering clinic sites,
* cannot identify a support person injector,
* has not received at least the loading dose of CAB/RPV,
* had serious adverse events with CAB/RPV with the loading dose,
* is not virologically suppressed,
* has a history of treatment failure,
* has a known or suspected resistance to either RPV or CAB,
* is not interested in receiving home-based injections,
* is not approved but their clinical team as a candidate for home-based injections;
* does not have the intention to use CAB/RPV for at least 12 months;
* and is not willing or unable to give informed consent.

Treatment Buddy:

* <18 years of age,
* is not willing or unable to provide monthly or bimonthly LAI-ART injections at the PWH's place of residence, and
* is not willing or unable to give informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: PWH who have been prescribed injectable cabotegravir/rilpivirine (CAB/RPV) as part of their routine care who have clinician approval to participate in the home-based program.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2026-02-16 (Estimated); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-09-29 (Estimated)

PRIMARY OUTCOMES:
Feasibility of Home-Based LAI-ART Administration | 12 months
  To assess Feasibility, HIV clinicians will complete the Feasibility of Intervention Measure. Possible scores on the Feasibility of Intervention Measure range from 4 (less feasible) to 20 (very feasible).
  Weiner BJ, Lewis CC, Stanick C, et al. Psychometric assessment of three newly developed implementation outcome measures. Implement Sci. 2017;12(1):108. Published 2017 Aug 29. doi:10.1186/s13012-017-0635-3
HIV viral suppression defined as two suppressed viral load test (HIV-RNA-PCR) results at least three months apart. | 12 months
  The investigators will assess viral suppression with two suppressed viral load test results at least three months apart within a 12-month period. A suppressed result is considered less than 200 copies/mL.

SECONDARY OUTCOMES:
Acceptability of Home-Based LAI-ART Administration | 12 months
  To assess Acceptability, People With HIV and their chosen Treatment Buddy will complete:
  1. Injection-Treatment Acceptance Questionnaire: Possible scores on the measure range from 0 (very unacceptable) to 120 (very acceptable).
  Tatlock S, Arbuckle R, Sanchez R, Grant L, Khan I, Manvelian G, Spertus JA. Psychometric Evaluation of a Treatment Acceptance Measure for Use in Patients Receiving Treatment via Subcutaneous Injection. Value Health. 2017 Mar;20(3):430-440. doi: 10.1016/j.jval.2016.09.2410. Epub 2016 Dec 1. PMID: 28292488.

CONTACTS AND LOCATIONS:
Overall Officials: Parya Saberi, PharmD, Principal Investigator — University of California, San Francisco
Locations (1):
- Division of Prevention Science, Center for AIDS Prevention Studies (CAPS), San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bourdeau B, Rebchook G, Shade SB, O'Shea J, Buchacz K, Harris O, Johnson MO, Palomares M, Bolton AT, Van Nuys J, Moore E, Saberi P. Innovative administration of long-acting injectables for HIV treatment enhancement at home (INVITE-HOME): implementation science study protocol. BMJ Open. 2025 Aug 5;15(8):e097921. doi: 10.1136/bmjopen-2024-097921. PMID 40764067